CLINICAL TRIAL: NCT05122637
Title: Feasibility Study of RapidPulseTM Aspiration System as Frontline Approach for Patients With Acute Ischemic Stroke Due to Large Vessel Occlusions
Brief Title: Feasibility Study of RapidPulseTM Aspiration System as Frontline Approach for Stroke Patients
Acronym: RapidPulseFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RapidPulse, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEV-0213
Record Dates: First submitted 2021-11-03; First posted 2021-11-17 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Acute Ischemic Stroke
Keywords: Large vessel occlusion; Mechanical thrombectomy; Neurovascular intervention
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): RapidPulseTM Aspiration System with commercially available Medtronic React 71 aspiration catheter and commercially available aspiration pump as frontline approach thrombectomy technique.
  Interventions: Device: RapidPulseTM Aspiration System
- Control Arm (Other): Treatment with commercially available aspiration catheter with commercially available aspiration pump as frontline approach thrombectomy technique.
  Interventions: Device: Standard of Care Aspiration Thrombectomy System

INTERVENTIONS:
Device: RapidPulseTM Aspiration System — The RapidPulseTM Aspiration System with Medtronic React 71 aspiration catheter and a commercially available pump.
  Arms: Treatment Arm
Device: Standard of Care Aspiration Thrombectomy System — Commercially available aspiration catheter with commercially available aspiration pump
  Arms: Control Arm

SUMMARY:
A Feasibility Study to evaluate the initial safety and performance of the RapidPulseTM Aspiration System in the treatment of patients with Acute Ischemic Stroke (AIS) due to Large Vessel Occlusion (LVO).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the initial safety and performance of the RapidPulse Inc. RapidPulseTM Aspiration System as frontline approach for use in the treatment of patients with Acute Ischemic Stroke (AIS) due to Large Vessel Occlusion (LVO). This is a prospective, multi-center, open label study comparing the safety and performance of the RapidPulseTM Aspiration System with non-randomized retrospective controls who otherwise meet the same study inclusion/exclusion criteria. The study will enroll a maximum of 100 participants in the Treatment Arm and a maximum of 200 participants in the Control Arm at in up to 10 centers in Europe and/or Latin America. Subjects data will be collected through hospitalization with a 3 months post-procedure study visit.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 years or older
* Clinical diagnosis of acute ischemic stroke with NIH Stroke Scale (NIHSS) score ≥ 6 with symptom onset (or last seen normal) up to 24 hours
* Large vessel occlusion in the intracranial internal carotid artery (ICA), middle cerebral artery (MCA) M1 or M2 segments, basilar or vertebral artery

Key Exclusion Criteria:

* Evidence of hemorrhage
* Significant mass effect and/or midline shift
* Vessel tortuosity too difficult to allow endovascular access per investigator judgment
* Severe or fatal co-morbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
First Pass Reperfusion Effect (FPE) | Intra-procedural
  Defined by modified Thrombolysis In Cerebral Infarction scale (mTICI 2c-3) flow in the target vessel

SECONDARY OUTCOMES:
Frontline technical success | Intra-procedural
  Defined by mTICI ≥ 2b after the last pass with Study Device with no rescue therapy
Good functional outcome measured by Modified Rankin Scale score of 0 - 2 at 90 days post index procedure | 90 days
  The Modified Rankin Scale (mRS) measures neurological disability or dependence for stroke patients on a scale of 0 (no symptoms) to 6 (deceased)
Rate of Symptomatic intracranial hemorrhage (sICH) at 24 hours post-procedure | 24 hours
All cause mortality rate | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Raul G Nogueira, MD, Study Chair — University of Pittsburgh Medical Center Stroke Institute
Locations (5):
- General Hospital of Fortaleza, Fortaleza, Brazil
- Odense University Hospital, Odense, Denmark
- Pauls Stradiņš Clinical University Hospital, Riga, Latvia
- Hospital General Universitari d'Alicante, Alicante, Spain
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No